CLINICAL TRIAL: NCT03435107
Title: A Phase II Study of Durvalumab in Patients With Mismatch Repair Deficient or POLE Mutated Metastatic Colorectal Cancer
Brief Title: Durvalumab for MSI-H or POLE Mutated Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Tae Won Kim, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-1151
Record Dates: First submitted 2018-02-07; First posted 2018-02-15 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab (Experimental): The mismatch repair deficient or microsatellite instable, or POLE mutated metastatic colorectal cancer patients who were refractory to fluoropyrimidines, irinotecan and oxaliplatin with or without targeted agents will be accrued.
  After checking the eligibility for the study entry, patients will be entered into the study treatment with durvalumab monotherapy.
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — Study treatment consists of durvalumab 1500 mg Q4W for patients > 30 kg, and will be repeated every 4 weeks. For patients ≤ 30 kg, weight based dosing of 20 mg/kg durvalumab Q4W will be used.
  Response evaluation will be performed every 8 weeks (± 1-week window period). Treatment will be continued until disease progression, unacceptable adverse events or the patient's refusal.
  Treatment through progression is at the investigator's discretion, and the investigator should ensure that patients do not have any significant, unacceptable, or irreversible toxicity that indicate that continuing treatment will not further benefit the patient. The Investigator should ensure that patients still meet all of the inclusion criteria and none of the exclusion criteria for this study.

SUMMARY:
The POLE mutations represent high somatic mutation loads in patients with colorectal cancer, especially in those with MMR proficient or MSS, therefore, tumors harbouring POLE mutations might be susceptible to immune checkpoint blockade.

Based on these reasons, the investigators planned a phase II study of durvalumab monotherapy in patients with previously treated, metastatic, MMR deficient (MSI-H) or POLE mutated colorectal cancer.

DETAILED DESCRIPTION:
Later-line therapies after failure of standard treatments for metastatic colorectal cancer patients are limited; regorafenib and TAS-102 have shown clinical activity for these patients, however, efficacy outcomes seemed not to be sufficient although there have been rather higher frequencies of adverse events.

Mismatch repair (MMR) deficiency or microsatellite instability-high (MSI-H) played a role of negative predictive factor for adjuvant fluorouracil-based chemotherapy in patients with resected colorectal cancer. In the metastatic setting, deficient MMR or MSI-H represented poor prognosis; however, their predictive role has been documented after the pembrolizumab trial was reported. The results of the pembrolizumab trial demonstrated that the PD-1 blockade with pembrolizumab monotherapy showed 40% of confirmed immune-related objective response rates in patients with MMR deficient metastatic colorectal cancers; hence there was no objective response in those with MMR proficient tumors. The progression-free rates at 20 weeks were 78% versus 11%, respectively, also favouring those with MMR deficient tumors. However, the MMR deficiency of MSI-H is found in only about 5% in patients with metastatic colorectal cancer, which is too small to expand potential candidate of immunotherapy.

One of the proposed mechanism of promising efficacy from pembrolizumab for MMR deficient colorectal cancer is that MMR deficient or MSI-H colorectal cancers harbour higher somatic mutation loads than MMR proficient colorectal cancer (a mean of 1782 somatic mutations per tumor in the MMR deficient tumors versus 73 in the MMR proficient tumors in the results of pembrolizumab trial); somatic mutations have the potential to encode non-self immunogenic antigens; therefore, immunotherapy enhancing immune surveillance produced promising treatment efficacy in the MMR deficient tumors.

The POLE gene encodes the catalytic subunit of DNA polymerase epsilon, and it involves DNA repair and chromosomal replication. The POLE mutations are located in the exonuclease domain, and their presence has already been reported in the various cancers including colorectal and endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed adenocarcinoma of the colon or the rectum.
2. Mismatch repair deficient or microsatellite instable (defined below), or POLE mutated tumors A. Mismatch repair deficient: loss of expression by immunohistochemical stains ≥ 1 out of 4 markers (MLH1, MSH2, MSH6, PMS2) B. Microsatellite instable: loss of stability ≥2 out of 5 gene panels (BAT-25, BAT-26, D2S123, D5S346, D17S250)
3. Refractory to at least one agent of prior treatments(fluoropyrimidines, irinotecan or oxaliplatin) Progressed after at least first-line systemic chemotherapy for metastatic setting (progressed within 6 months after completion of adjuvant chemotherapy is also considered as first-line failure)
4. ≥ 1 measurable lesion(s) by RECIST 1.1.
5. Unresectable advanced or metastatic disease.
6. Age over 20 years old.
7. ECOG performance status of 0-1 or lower.
8. Adequate organ functions. A. Bone marrow function: Hemoglobin 9.0≥ g/dL, ANC≥ 1,500/mm3, platelet≥ 100,000/mm3 B. Hepatic functions: bilirubin ≤ 1.5 X ULN, AST/ALT ≤ 2.5 X ULN (≤ 5 X ULN in cases of liver metastasis) C. Renal functions: serum Cr ≤ 1.5 X ULN or calculated CCr (Cockcroft) > 40 ml/min
9. Be willing and able to comply with the protocol for the duration of the study.
10. Give written informed consent prior to study-specific screening procedures, with the understanding that the patient has the right to withdraw the study at any time, without prejudice.
11. Female subjects must either be of non-reproductive potential (≥ 60 years old and no menses for ≥ 1 year without an alternative medical cause, or history of hysterectomy, or history of bilateral tubal ligation, or history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.
12. Women of childbearing potential and men must agree to use adequate contraception since signing of the IC form until at least 90days after the last study drug administration.

Exclusion Criteria:

1. Any prior treatment with PD-1 or PD-L1 inhibitor, including durvalumab.
2. Involvement in the planning and/or conduct of the study.
3. Receipt of the last dose of chemotherapy ≤ 28 days prior to the first dose of study drugs.
4. Mean QT interval corrected for heart rate (QTc) ≥ 470 msec calculated from 3 electrocardiograms (ECGs) using Frediricia's Correction.
5. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria
6. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
7. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
8. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (eg, hormone replacement therapy) is acceptable.
9. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiologic doses, which are not to exceed 10 mg/day of prednisolone, or an equivalent corticosteroid.
10. Concurrent or previous history of another primary cancer within 3 years prior to randomisation except for curatively treated cervical cancer in situ, non-melanomatous skin cancer, superficial bladder cancer (pTis and pT1) and curatively treated thyroid cancer of any stage. Concurrent, histologically confirmed, unresected thyroid cancer without distant metastasis could be allowed with the agreement of the chief principal investigator.
11. Uncontrolled CNS metastases; permitted if asymptomatic or neurologically stable.
12. Prior radiation therapy would be permitted, but non-radiated evaluable lesions should be present at study entry.
13. Radiation therapy during study treatment is not permitted, but if the local investigator decides that radiation therapy should be given during study treatments, he should be convinced that there is no evidence of disease progression with agreement of the chief principal investigator.
14. Congestive heart failure ≥ New York Heart Association (NYHA) class 2.
15. Unstable angina, new-onset angina within 3 months, or history of myocardial infarction within 6 months before the study entry.
16. Active or prior documented autoimmune disease within the past 2 years; subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
17. Active or prior documented inflammatory bowel disease.
18. History of prior immunodeficiency.
19. History of allogeneic organ transplantation.
20. History of hypersensitivity to durvalumab or any excipient.
21. History of previous clinical diagnosis of active tuberculosis.
22. Receipt of live attenuated vaccination within 30 days prior to study entry.
23. Known history of testing positive for HIV
24. Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive) Except, resolved HBV infection (as evidenced by detectable HBV surface antibody, detectable HBV core antibody, undetectable HBV DNA, and undetectable HBV surface antigen) or Chronic HBV infection (as evidenced by detectable HBV surface antigen or HBV DNA). Subjects with chronic HBV infection must have HBV DNA < 100 IU/mL and must be on antiviral therapy.
25. Major surgery or significant traumatic injury within 28 days prior to study treatment.
26. Non-healing wound, ulcer, or bone fracture.
27. Current evidence of significant gastrointestinal bleeding or (impending) obstruction.
28. Concomitant participation in another clinical trial.
29. Pregnant of breast-feeding subjects. Women of child-bearing potential must have pregnancy test within 7 days and a negative result must be documented before start of study treatment.
30. Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tae Won Kim, Professor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Durvalumab: The mismatch repair deficient or microsatellite instable, or POLE mutated metastatic colorectal cancer patients who were refractory to fluoropyrimidines, irinotecan and oxaliplatin with or without targeted agents will be accrued.
  After checking the eligibility for the study entry, patients will be entered into the study treatment with durvalumab monotherapy.
  Durvalumab: Study treatment consists of durvalumab 1500 mg Q4W for patients > 30 kg, and will be repeated every 4 weeks. For patients ≤ 30 kg, weight based dosing of 20 mg/kg durvalumab Q4W will be used.
  Response evaluation will be performed every 8 weeks (± 1-week window period). Treatment will be continued until disease progression, unacceptable adverse events or the patient's refusal.
  Treatment through progression is at the investigator's discretion, and the investigator should ensure that patients do not have any significant, unacceptable, or irreversible toxicity that indicate that continuing treatment will not further benefit the patient. The Investigator should ensure that patients still meet all of the inclusion criteria and none of the exclusion criteria for this study.
Period: Overall Study
Arm/Group | Durvalumab
Started | 33
Completed | 32
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Durvalumab
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 33
Region of Enrollment [Number; unit: participants]
  South Korea | 33
Primary tumor [Count of Participants; unit: Participants]
  Right colon | 21
  Left colon | 9
  Rectum | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rates (RECIST 1.1)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI:
  Complete Response (CR): Disappearance of all target lesions Partial Response (PR):>=30% decrease in the sum of the longest diameter of target lesions Overall Response (OR) = CR + PR
Time Frame: First measurement should be at 8weeks from first administration.After first measurement, it should be followed up at every 8weeks until date of progression disease or date of death from any cause, whichever came first, assessed up to 46months..
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Durvalumab
Number analyzed (Participants) | 33
Percentage of participants | 42.4 [25.5 to 60.8]

2. Secondary Outcome: Disease Control Rate (DCR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI:
  Disease control rate (DCR); The percentage of patients with the best overall response of complete response (CR), partial response (PR), or stable disease (SD) sustained for at least 6 weeks.
Time Frame: Through study completion, an average of 2 years and 3months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Durvalumab
Number analyzed (Participants) | 33
Percentage of participants | 66.7 [48.2 to 82.0]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected through study treatment completion, an average of 1 year and 4months. All-Cause Mortality was assessed up to 46months
Description: The term adverse event covers any unfavorable and unintended sign, symptom, syndrome, or illness that develops or worsens during the period of observation in the clinical study.
Arm/Group | Durvalumab
All-Cause Mortality (participants affected / at risk) | 15/33
Serious Adverse Events (participants affected / at risk) | 13/33
Other Adverse Events (participants affected / at risk) | 28/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab (N=33)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Infection (Infections and infestations) | 1
Acute Kidney Injury (Renal and urinary disorders) | 2
Both knee pain (Musculoskeletal and connective tissue disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Atypical ductal hyperplasia of breast (Reproductive system and breast disorders) | 1
Anal fistula (Skin and subcutaneous tissue disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Durvalumab (N=33)
Hyperthyroidism (Endocrine disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Serum sickness-like reaction (Immune system disorders) | 1
Neutrophil count decreased (Investigations) | 1
Anemia (Investigations) | 4
Platelet count decreased (Investigations) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 8
Fatigue (General disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 5
Oral mucositis (Skin and subcutaneous tissue disorders) | 5
Increased lipase (Investigations) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Diarrhea (Gastrointestinal disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Aspartate aminotransferase increased (Investigations) | 3
Alanine aminotransferase increased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 2
Increased amylase (Investigations) | 2
Nausea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Dizziness (Nervous system disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 2
Hypothyroidism (Endocrine disorders) | 5
Thromboembolism (Vascular disorders) | 1
White blood cell decreased (Investigations) | 1
Pancreatitis (Gastrointestinal disorders) | 2
Skin rash (Skin and subcutaneous tissue disorders) | 3
Acute kidney injury (Renal and urinary disorders) | 3
Peripheral edema (General disorders) | 3
Peripheral neuropathy (Nervous system disorders) | 3
Hypercholesterolemia (Metabolism and nutrition disorders) | 2

LIMITATIONS AND CAVEATS:
The limitations of the present study include a relatively small sample size, the absence of a control group and a short follow-up duration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/07/NCT03435107/Prot_SAP_000.pdf